CLINICAL TRIAL: NCT05094830
Title: Stomach Intestinal Pylorus Sparing (SIPS) As a Primary and Revisional Bariatric Surgery
Brief Title: Stomach Intestinal Pylorus-Sparing Bariatric Surgery
Acronym: SIPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment barriers
Sponsor: Bradley Needleman (Other)
Responsible Party: Sponsor-Investigator, Bradley Needleman, Professor of Surgery, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017H0400
Record Dates: First submitted 2018-05-23; First posted 2021-10-26 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2023-10

CONDITIONS: Obesity
Keywords: Weight Loss Surgery; Bariatric Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stomach Intestinal Pylorus Sparing (SIPS) (Experimental): Patients undergoing SIPS procedure as their bariatric surgery of choice.
  Interventions: Procedure: Stomach Intestinal Pylorus-Sparing (SIPS) Procedure

INTERVENTIONS:
Procedure: Stomach Intestinal Pylorus-Sparing (SIPS) Procedure — The SIPS procedure will be performed as an investigational bariatric surgery. The SIPS procedure involves the creation of a standard sleeve gastrectomy over a 36-40 bougie. Division of the duodenum post-pylorus is performed, followed by the creation of a common channel 300 cm from the ileo-cecal valve. A hand-sewn anti-side duodenoileostomy is performed and the anastomosis tested for leaks through use of endoscopic insufflation and under water air leak test. Incisions are then closed in standard fashion. The SIPS procedure itself is not a separate surgery but rather a modification to the standard of care surgery.

SUMMARY:
This study will evaluate the safety and efficacy of Stomach Intestinal Pylorus Sparing (SIPS) as a primary bariatric surgery. In addition, we will evaluate the safety and efficacy of SIPS performed as a revisional surgery following sleeve gastrectomy (SG) in which adequate weight loss was not achieved.

DETAILED DESCRIPTION:
This is a prospective study of an interventional procedure. Results of patients selecting to undergo the Stomach Intestinal Pylorus Sparing (SIPS) procedure will be prospectively collected.

In addition to the currently offered bariatric weight loss procedures, patients who present to our bariatric clinic will be presented with information on the SIPS procedure. All patients interested in pursuing bariatric surgery will undergo a standardized bariatric surgery evaluation process as standard of care. Patients interested in undergoing SIPS must meet the following inclusion/exclusion criteria in addition to the established criteria for bariatric surgery.

The SIPS procedure will be performed as an investigational procedure. The SIPS procedure involves the creation of a standard sleeve gastrectomy over a 36-40 bougie. Division of the duodenum post-pylorus is performed, followed by the creation of a common channel 300 cm from the ileo-cecal valve. A hand-sewn anti-side duodenoileostomy is performed and the anastomosis tested for leaks through use of endoscopic insufflation and under water air leak test. Incisions are then closed in standard fashion. The SIPS procedure itself is not a separate surgery but rather a modification to the standard of care surgery.

All patients electing to enroll in this study will experience the same pre- and postoperative care provided as standard of care to all bariatric surgery patients. A pre-operative evaluation is performed to confirm appropriateness for bariatric surgery and includes: Psychological evaluation, dietary counseling, and testing of cardiovascular, pulmonary, and gastrointestinal health. Pre-operative evaluation also consists of blood work to identify or confirm obesity-related comorbid conditions. Post-operative care provided following bariatric surgery ensures that patients progress with adequate pain control and appropriate diet tolerance before hospital discharge while evaluating and monitoring manifestations of potential complications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-89
* Primary: Satisfies established NIH criteria for bariatric surgery
* Revision of sleeve gastrectomy: Sleeve gastrectomy performed at least two years prior but the patient did not reach 50% excess weight loss (EWL), has regained 20% of EWL since sleeve gastrectomy, or has current BMI > 40
* Willing and able to provide his/her own consent for the surgery

Exclusion Criteria:

* Contraindication to bariatric surgery
* Current pregnancy/breast feeding or plans for pregnancy
* Prisoners
* Previous history of gastrectomy other than sleeve gastrectomy for weight loss
* History of small bowel resection
* History of any kind of surgery to treat gastroesophageal reflux disease (GERD)
* History of or current Barrett's esophagus
* History of or any kind of cancer diagnosis in last 5 years
* Large hiatal hernia > 5 cm

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Safety as a primary procedure | Short-term (30 days)
  Complication rates
Efficacy as a primary procedure | Long-term (5 years)
  Excess weight loss achieved post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Needleman, MD, Principal Investigator — The Ohio State University College of Medicine
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No